CLINICAL TRIAL: NCT02247661
Title: Hip Abductor Strengths, Limping and Trochanteric Tenderness After Hip Arthroplasty Due to Femoral Neck Fracture: A Comparison Between the Lateral and Posterolateral Approaches
Brief Title: Hip Abductor Strengths, Limping and Trochanteric Tenderness After Hip Arthroplasty Due to Femoral Neck Fracture
Acronym: HASAP
Status: Completed | Type: Observational
Sponsor: Sundsvall Hospital (Other)
Responsible Party: Principal Investigator, Lennart Bråbäck, Head FoU, Sundsvall Hospital
Other Study IDs: SM_II
Record Dates: First submitted 2014-09-20; First posted 2014-09-25 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Femoral Neck Fracture; Trochanteric Pain
Keywords: Femoral neck fracture,surgical approach, limp, abductor strenght, trochanteric pain
MeSH Terms: conditions — Femoral Neck Fractures; Intermittent Claudication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Direct lateral approach: Total or hemiarthroplasty operated with direct-lateral approach.
- Postero-lateral approach: Total or hemiarthroplasty operated with postero-lateral approach.

SUMMARY:
A prospective cohort study to compare the direct lateral and poster-lateral approach concerning abductor function. Patients admitted with a femoral neck fracture operated with a hemiarthroplasty through a direct lateral or a poster-lateral approach were screened for inclusion. Patients with altered mental status SPMSQ >7, pathological fractures, non-walkers were excluded.

Those who fulfilled the inclusion criteria and non of the exclusion criteria were followed 1 year postoperatively by clinical examination. Sample size were estimated to 30 patient in each group. Primary outcome variables were trendelenburg test, abductor strength measured with dynamometry, trochanteric tenderness measured with algometry and palptation.

ELIGIBILITY:
Inclusion Criteria:

* Displaced femoral neck fracture
* Walker
* Hemarthroplasty
* Preiffer test >7/10

Exclusion Criteria:

* Pathological fracture
* Non-walker
* Pfeiffer test <7/10 indicating mental alteration.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Sundsvall hospital with a displaced femoral neck fracture operated with either a total or hemiarthroplasty.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Trendelenburg Test | 1 year
  30 seconds standing on the operated leg

SECONDARY OUTCOMES:
Abductor strenght | 1 year
  Dynamometry
Trochanteric tenderness | 1 year
  Algometry
Trochanteric tenderness | 1 year
  Palptation

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopaedic department, Sundsvall hospital, Sundsvall, Västernorrland County, Sweden

REFERENCES:
- [Background] Skoldenberg O, Ekman A, Salemyr M, Boden H. Reduced dislocation rate after hip arthroplasty for femoral neck fractures when changing from posterolateral to anterolateral approach. Acta Orthop. 2010 Oct;81(5):583-7. doi: 10.3109/17453674.2010.519170. PMID 20860452
- [Background] Pai VS. Significance of the Trendelenburg test in total hip arthroplasty. Influence of lateral approaches. J Arthroplasty. 1996 Feb;11(2):174-9. doi: 10.1016/s0883-5403(05)80013-0. PMID 8648312
- [Background] Kiyama T, Naito M, Shinoda T, Maeyama A. Hip abductor strengths after total hip arthroplasty via the lateral and posterolateral approaches. J Arthroplasty. 2010 Jan;25(1):76-80. doi: 10.1016/j.arth.2008.11.001. Epub 2009 Apr 8. PMID 19359133